CLINICAL TRIAL: NCT03321110
Title: Effects of Coenzyme Q10 Supplementation on Oxidative Stress, Antioxidant Capacity, Inflammatory Responses, Fatigue Elimination, and Exercise Performance in Athletes From Different Sports: Cross-sectional, Interventional, and Follow-up Studies
Brief Title: Effects of Coenzyme Q10 Supplementation on Oxidative Stress, Antioxidant Capacity, Inflammatory Responses, Fatigue Elimination, and Exercise Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, LJ Hwu, Principal Investigator, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MOST106-2410-H-030-065
Record Dates: First submitted 2017-10-13; First posted 2017-10-25 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Athlete
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: placebo-control
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): Placebo
  Interventions: Other: Placebo
- Q10-150 (Experimental): coenzyme Q10 150 mg/d.
  Interventions: Dietary Supplement: Coenzyme Q10
- Q10-300 (Experimental): coenzyme Q10 300 mg/d.
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Other: Placebo — Placebo (dextrin)
  Arms: Placebo
Dietary Supplement: Coenzyme Q10 — 150 mg or 300 mg
  Arms: Q10-150; Q10-300

SUMMARY:
The aims of the study are 1) to compare the differences in plasma coenzyme Q10, oxidative stress, antioxidant capacity, muscle impairment, fatigue recovery, and inflammation and exercise performances in athletes (i.e., soccer, and taekwondo players) and healthy non-athletes; 2) to investigate the relationship between plasma coenzyme Q10, oxidative stress, antioxidant capacity, muscle impairment, fatigue recovery, and inflammation and exercise performances; 3) to explore the influence on plasma coenzyme Q10, oxidative stress, antioxidant capacity, muscle impairment, fatigue recovery, and inflammation and exercise performances after 12 weeks of coenzyme Q10 intervention (150 mg/day and 300 mg/day).

DETAILED DESCRIPTION:
The long-term high-amount and -intensity exercise training could cause oxidative damage, muscle impairment, inflammation and exercise fatigue to athletes easily. Such above conditions will affect the exercise performances and health of athletes. The aims of the study are 1) to compare the differences in plasma coenzyme Q10, oxidative stress, antioxidant capacity, muscle impairment, fatigue recovery, and inflammation and exercise performances in athletes (i.e., soccer, and taekwondo players) and healthy non-athletes; 2) to investigate the relationship between plasma coenzyme Q10, oxidative stress, antioxidant capacity, muscle impairment, fatigue recovery, and inflammation and exercise performances; 3) to explore the influence on plasma coenzyme Q10, oxidative stress, antioxidant capacity, muscle impairment, fatigue recovery, and inflammation and exercise performances after 12 weeks of coenzyme Q10 intervention (150 mg/day and 300 mg/day). Eventually, these results of this study can provide the information for the known to improve the oxidative stress, anti-oxidation and inflammation internal to the bodies of athletes for various competitions. As a consequence, the athletic performances can be further enhanced.

ELIGIBILITY:
Inclusion Criteria:

* Athletes (soccer and taekwondo players)

Exclusion Criteria:

* Antioxidant vitamins users
* Statins or Aspirin therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
malondialdehyde (MDA) | 12 weeks
  MDA (micromol/L) will measure by thiobarbituric acid reacting substance.

SECONDARY OUTCOMES:
Antioxidant capacity | 12 weeks
  Total antioxidant capacity (TAC) was measured by a Trolox equivalent antioxidant capacity assay in serum and erythrocytes.
high sensitivity C-reactive protein (hs-CRP) | 12 weeks
  hs-CRP will measure by immunoturbidimetry.
creatine kinase (CK) | 12 weeks
  serum CK will measure by enzymatic method.
Lactate dehydrogenase (LDH) | 12 weeks
  serum LDH will measure by enzymatic method.
one-repetition maximum (1-RM) | 12 weeks
  1RM measurements will report in kilograms for data analysis.
Glucose | 12 weeks
  mmol/L
HbA1C | 12 weeks
  HbA1C will measure by an automated glycated hemoglobin analyzer
Insulin | 12 weeks
  insulin will measure by an automated chemistry analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No